CLINICAL TRIAL: NCT05183841
Title: Effect of Bronchodilators on the Exercise Capacity of Bronchiectasis Patients
Brief Title: Bronchodilators on the Exercise Capacity of Bronchiectasis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Celso R. Carvalho, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3008.886
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Bronchiectasis Adult
Keywords: Bronchiectasis; Bronchodilators Agents; Exercise/Physical Activity; Respiratory Mechanics
MeSH Terms: conditions — Bronchiectasis; Motor Activity | interventions — Bronchodilator Agents; Ipratropium; Fenoterol; fenoterol, ipratropium drug combination

STUDY DESIGN:
Intervention Model Description: On the first day, anamnesis, anthropometric evaluation and lung function will be performed, followed by: Quality of Life Questionnaire-Bronchiectasis, Saint George questionnaire, modified Medical Research Council scale and social and economic status. Then, a cardiopulmonary exercise test (CPET) will be performed and after rest, a bronchodilator (BD) or placebo randomization will precede a constant load exercise test (CLET) with the respiratory mechanics assessment (OEP). Finally, the accelerometer will be coupled to the patient for 7 consecutive days, aiming to assess the PAL. On the second day, after at least one-week washout, the accelerometer will be collected and the patient will repeat the CLET with the respiratory mechanics assessment, at the opposite condition to randomization.
Who Masked: Participant, Outcomes Assessor
Masking Description: All the measurements will be performed by a blinded professional, who will be masked from randomization and other results. The randomization sequence will be generated by computer, and put in sealed and opaque envelopes by a volunteer not involved in the study. The bronchodilator (BD) or placebo will be administered by a professional not involved in the study, according to the randomization. The evaluator will not have access to information on which intervention (BD or placebo) was given prior to each CLET.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bronchodilator (Active Comparator): The intervention will be a combination of 2 drugs, ipratropium (20 mcg) and fenoterol (50mcg). Ipratropium is an anticholinergic bronchodilator, and fenoterol is a beta-agonist bronchodilator. The medication will be delivered to the patient via an inhaler device with spacer, at leat 20 minutes before the constant load exercise test (CLET). Patient will be asked for a total exhalation, followed by an appropriate spacer mouthpiece placement and the first of eight puffs (30 seconds interval between puffs) will be delivered through the opposite extremity of the spacer. Patient will be instructed to perform five tidal volume breaths for each puff.
  Interventions: Drug: Bronchodilator (Ipratropium and Fenoterol)
- Placebo (Placebo Comparator): The placebo will be delivered via an inhaler device with spacer (identical to the bronchodilator device), at least 20 minutes before the constant load exercise test (CLET). Patient will be asked for a total exhalation, followed by an appropriate spacer mouthpiece placement and the first of eight puffs (30 seconds interval between puffs) will be delivered through the opposite extremity of the spacer. Patient will be instructed to perform five tidal volume breaths for each puff.
  Interventions: Other: Placebo
- Control (No Intervention): A paired healthy control group will be assessed by a constant load exercise test (75% from maximal load achieved on the cardiopulmonary exercise test) concomitant to the optoelectronic plethysmography to compare mechanical respiratory parameters to the bronchiectasis patients during the placebo assessment. In addition they will also use an accelerometer for 7 consecutive days.

INTERVENTIONS:
Drug: Bronchodilator (Ipratropium and Fenoterol) — 8 puffs of Ipratropium (20mcg) and Fenoterol (50mcg) via an inhaler device with a spacer (30 seconds interval between puffs) in 5 tidal volume breaths each puff.
  Other Names: duovent
  Arms: Bronchodilator
Other: Placebo — 8 puffs of placebo via an inhaler device with a spacer (30 seconds interval between puffs) in 5 tidal volume breaths each puff.
  Arms: Placebo

SUMMARY:
The bronchodilators (BD) have been widely used in bronchiectasis (BCE) therapeutic and have been shown to be effective in improving exercise capacity in patients with chronic obstructive pulmonary disease and asthma. However the BD effect on the exercise capacity of patients with BCE is poorly known. Besides, the respiratory mechanics pattern of the patients with BCE is not known nor its association with their physical activity level (PAL). Therefore, the hypothesis of this study is that BD are effective in improving exercise capacity of patients with BCE. The authors also propose to characterize the respiratory mechanics of the patients with BCE and to evaluate their PAL and its association with quality of life, as secondary aims.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover, placebo-controlled trial. Forty clinically stable patients with bronchiectasis (BCE), all sexes, 18 to 59 years, will be evaluated in two non-consecutive days. On the first day, anamnesis, anthropometric evaluation and lung function will be performed, followed by: Quality of Life Questionnaire-Bronchiectasis, Saint George questionnaire, modified Medical Research Council scale and social and economic status. Then, a cardiopulmonary exercise test (CPET) will be performed and after a rest period, a bronchodilator (BD) or placebo randomization will precede a constant load exercise test (CLET) with the respiratory mechanics assessment (OEP). Spirometry will be performed pre and post BD/placebo. Finally, the accelerometer will be coupled to the patient for 7 consecutive days, aiming to assess the PAL. On the second day, after at least one-week washout, the accelerometer will be collected and the patient will repeat the CLET with the respiratory mechanics assessment, at the opposite condition to the randomization. The randomization sequence will be generated by computer, and put in sealed and opaque envelopes by a volunteer not involved in the study. The BD or placebo will be administered by a volunteer not involved in the study, according to the randomization. The evaluator will not have access to information on which intervention (BD or placebo) was given prior to each CLET. A paired (anthropometric and social and economic status) healthy control group will be assessed by spirometry, CPET, and CLET and OEP, for comparing respiratory mechanics. In addition the participants will also use an accelerometer for 7 consecutive days. Data of endurance time from CLET, respiratory mechanics from OEP, dyspnea and vital signs will be assessed before and after both BD and placebo CLET. Data about onset of BCE, comorbidities and BCE medication will be collected from the patient's medical record. Data normality will be tested by Kolmogorov-Smirnov. Data comparison will be performed by t test or Wilcoxon and the association by Pearson or Spearman. Categorical data will be analyzed by qui-square test or Fischer. The significance level will be set to 5% for all tests.

ELIGIBILITY:
Inclusion Criteria:

* All sexes
* 18 to 59 years
* Bronchiectasis diagnosis, according to thorax the Computed Tomography (Pasteur et al., 2010)
* Clinically stable (last 30 days without exacerbation/hospitalization)
* Air trapping on plethysmography (Residual Volume/Total Lung Capacity>125%)
* Smoking Load <10 pack-years

Exclusion Criteria:

* Do not accept to participate
* Smoking
* Continuous oxygen use
* Pulmonary Rehabilitation program in the last 6 months
* Previous lung resection
* Uncontrolled cardiovascular disease
* Other respiratory chronic diseases
* Neurological or musculoskeletal disorders that limit exercise
* Cognitive deficits that limit comprehension

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
endurance time | 60 seconds
  Endurance time will be assessed by the constant load exercise test (CLET). The CLET will be performed with 75% of maximal load (W) achieved on the cardiopulmonary exercise test (CPET). The CLET will be performed at a cycloergometer and the end of the CLET will be determined by the exertion (modified Borg Scale 9-10) or the required pedaling rate (60/min.) could not be kept up for 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Director — University of São Paulo General Hospital
Locations (3):
- Brazil (3):
  - Celso Ricardo Fernandes de Carvalho, São Paulo
  - Clinical Hospital of Sao Paulo University Medical School (HCFMUSP), São Paulo
  - Clinical Hospital of Sao Paulo University Medical School, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques da Silva CCB, Dal Corso S, Lunardi AC, Fonseca AJ, Rached SZ, Athanazio RA, Carvalho CRF. Effect of Dual Bronchodilation on the Exercise Capacity of Individuals With Non-Cystic Fibrosis Bronchiectasis: Protocol for a Randomized Controlled Double-Blind Crossover Study. JMIR Res Protoc. 2025 Jul 28;14:e68582. doi: 10.2196/68582. PMID 40720815